CLINICAL TRIAL: NCT03606304
Title: Using Problem-solving Intervention (PST-HF) to Improve Depressive Symptoms and Self- Care Ability Among Recently Hospitalized Older Patients With Heart Failure: A Feasibility Study
Brief Title: Problem-solving to Improve Depressive Symptoms and Self- Care Among Recently Hospitalized Adults With Heart Failure
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: The study was not deemed feasible to conduct.
Sponsor: University of Rochester (Other)
Responsible Party: Principal Investigator, Jinjiao Wang, Assistant Professor, University of Rochester
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SON2018-002
Record Dates: First submitted 2018-07-17; First posted 2018-07-30 (Actual); Last update posted 2019-07-08 (Actual); Status verified 2019-07

CONDITIONS: Heart Failure; Depression
Keywords: self-care; quality of life
MeSH Terms: conditions — Heart Failure; Depression

STUDY DESIGN:
Intervention Model Description: This is a single group, pre-/post-test design with a 6 month follow-up period. There are 8 weekly intervention sessions, each approximately 30-45 minutes long. The 3 telephone booster sessions occurring every two months during the followup phase are estimated to last 20 minutes.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Problem-solving therapy (Experimental): The intervention is based on an established PST protocol for medical patients, with an additional focus on HF to link depressed mood to impaired HF self-care. Seven steps are included: 1) select and define the problem; 2) establish realistic and achievable goals for problem resolutions; 3) generate multiple solution alternatives (brainstorming); 4) implement decision-making guidelines (pros and cons); 5) evaluate and choose the solutions; 6) implement the preferred solution(s); and 7) evaluate the outcome.
  Interventions: Behavioral: Problem-solving therapy

INTERVENTIONS:
Behavioral: Problem-solving therapy — See previous

SUMMARY:
The purpose of this study is to examine the feasibility of providing a problem-solving therapy-based intervention to improve both depressive symptoms and heart failure self-care specifically after hospital discharge. This is because the period after hospital discharge is critical to long-term recovery, overall quality of life, and prevention of adverse outcomes, such as hospital readmission.

DETAILED DESCRIPTION:
Depressive symptoms and impaired self-care respectively occur in up to 58% and 80% of older hospitalized patients with heart failure, and each doubles the risk of rehospitalization. These two conditions are closely intertwined with shared core behaviors/experiences, i.e., hopelessness/negative expectation, loss of motivation, impaired problem-solving skills, and social isolation/poor social support. As such, integrated interventions that explicitly address both depressive symptoms and impaired HF self-care are more efficacious than interventions that focus on depressive symptoms or HF self-care alone. In separate studies, problem-solving therapy (PST) has been effective to improve depressive symptoms and self-care for heart disease in older adults, including those with mild cognitive impairment. Though promising, there is no evidence regarding PST efficacy in addressing both depressive symptoms and self-care in HF patients. This is due to 1) sample heterogeneity, as only 18% to 77% of the subjects in prior studies had HF, and 2) separate interventional foci, as HF information was not used to link depressed mood to impaired self-care. Characteristics of hospitalized HF patients such as timing and cognitive function were also not considered. The first three months after hospital discharge is the period when depressive symptoms are most likely to change and when impaired HF self-care is mostly likely to lead to rehospitalization. Moreover, more than half (54%) of older depressed HF patients have mild cognitive impairment that can lead to dementia, especially in the context of impaired self-care, uncontrolled HF and restricted cerebral blood flow. However, no PST interventions have been specifically provided in the post-discharge period or among HF patients with mild cognitive impairment. To date, there is no evidence regarding the efficacy of integrated PST interventions on both depressive symptoms and impaired self-care in HF patients after hospital discharge.

The ultimate goal of this research program is to prevent rehospitalization in HF patients using integrated PST interventions to simultaneously improve depressive symptoms and self-care. Built on the investigator's prior work with depressive symptoms in home health care (HHC), this study will examine the feasibility of a home-based, telephone-enhanced PST intervention (PST-HF) in these patients after hospital discharge.

ELIGIBILITY:
Inclusion Criteria:

1. age ≥ 65;
2. having a primary diagnosis of HF (New York Heart Association [NYHA] Class I, II, III) of the index hospitalization;
3. having clinically significant depressive symptoms (PHQ-9 score≥10) at both hospital discharge and four weeks after hospital discharge;
4. inadequate HF self-care ability (any domain score in the Self-Care of Heart Failure Index [SCHFI]≤70/100); and
5. having normal or mildly impaired cognitive function (score of Montreal Cognitive Assessment [MoCA]: 23-30).

Exclusion Criteria:

1. being listed for an implanted ventricular assist device, heart transplant or currently receiving Milrinone infusion (indicating decompensated HF);
2. receiving hospice care or end-of-life care;
3. having diagnoses of the following, a) delirium or advanced Alzheimer's disease, b) malignant cancer, coronary artery disease requiring surgery or angioplasty, renal disease on dialysis in the present or within the past two years, c) severe psychotic disorder or suicidal ideation (or scored "0" in PHQ-9 item #9);
4. initiation or titration of antidepressants in the past 8 weeks; or
5. inability to give informed consent and/or to communicate verbally in English.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-05 (Estimated); Primary Completion 2019-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Problem-solving skills | 6 months post-discharge
  problem solving skills as measured by the Social Problem-Solving Inventory-Revised (Short) SPSI-R:S: There are 25 items measuring 5 components: Positive Problem Orientation, Negative Problem Orientation, Rational Problem Solving, Impulsivity/Carelessness Style, and Avoidance Style. Validated norms are provided by age group and raw scores are plotted for conversion to standard scores. Higher scores reflect greater intensity of the construct measured.

SECONDARY OUTCOMES:
Behavioral Activation for Depression | 6 months post-discharge
  Behavioral activation as measured by the Behavioral Activation for Depression Scale-Short Form (BADS-SF): ( item instrument with scores ranging from 0=not at all to 6=completely. Item scores are summed and higher scores indicate increased activation.
Depressive symptoms | 6 months post-discharge
  Depressive symptoms as measured by the Patient Health Questionnaire-9 (PHQ-9): 9 items with item anchors of 0=Not at all to 3=nearly every day; scale scores range from 0-27 with higher scores indicating greater depressive symptoms
Depressive symptoms | 6 months post-discharge
  Depressive symptoms as measured by the Hamilton Depression Rating Scale (HAM-D): Scores are based on 17 items with higher scores indicative or higher depressive symptoms. Scores 0-7 are classified as "normal"; 8-13="mild depression"; 14-18="moderate depression"; 19-22="severe depression; and >=23="very severe depression"
Heart Failure Self-care | 6 months post-discharge
  Heart failure self-care as measured by the Self-Care of Heart Failure Index (SCHFI): There are 3 scales: Self-Care Maintenance, Self-Care Management, and Self-Care Confidence. Self-Care Maintenance (10 items) assess self-care behaviors and each item is scored from 1=Never/rarely to 4=Always/daily. The Self-Care Management scale has 7 items. Item #11 is scored from 0=I did not recognize it to 4=Very quickly; item #s12-15 are scored from 1=Not likely to 4=Very likely; and item #16 is scored from 0=I did not try anything to 4=Very sure. The Self-Care Confidence scale has 6 items scored from 1=not confident to 4=extremely confident. All scales scores are standardized yileding scores ranging from 0 to 100.

CONTACTS AND LOCATIONS:
Overall Officials: Tiffany Gommel, MS, CIM, CIP, Study Director — University of Rochester

IPD SHARING:
Plan to Share IPD: No